CLINICAL TRIAL: NCT02916511
Title: Study of Extensive Clinical Target Volumes in Postoperative Radiotherapy Concurrent With Chemotherapy for Esophageal Squamous Cell Carcinoma
Acronym: ESO-Shanghai9
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Kuai Le Zhao, MD, Professor, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ESO-Shanghai9
Record Dates: First submitted 2016-09-26; First posted 2016-09-27 (Estimated); Last update posted 2023-12-22 (Actual); Status verified 2023-12

CONDITIONS: Esophageal Squamous Cell Carcinoma
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — Paclitaxel; Carboplatin; Radiotherapy

ARMS (1):
- Chemo-radiation group (Experimental): A total dose of 45Gy will be delivered in 25 fractions at 1.8Gy/fraction, 5 fractions per week in 5 weeks.
  The CTV encompassed the bilateral supraclavicular region, all mediastinal lymph nodes, the anastomosis site, and the left gastric and celiac nodes.
  Paclitaxel 50mg/m2/d, ivgtt over 3 hours, d1; Carboplatin AUC=2, ivgtt, d1; qw*5
  Interventions: Drug: Paclitaxel; Drug: Carboplatin; Radiation: Radiotherapy

INTERVENTIONS:
Drug: Paclitaxel — paclitaxel 50mg/m2/d, ivgtt over 3 hours, d1, qw*5
Drug: Carboplatin — carboplatin AUC=2, ivgtt, d1, qw*5
Radiation: Radiotherapy — 1.8Gy/d, d1-5/week, 25Fx

SUMMARY:
The purpose of this study is to evaluate safety and 2-year local control rate for extensive clinical target volumes in postoperative radiotherapy concurrent with chemotherapy for esophageal squamous cell carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Joined the study voluntarily and signed informed consent form;
* Age 18-75;
* ECOG 0-2;
* Esophageal squamous cell carcinoma, radical surgery ≤ 3 months, R0 resection;
* The operative incision healed well;
* T3-4N0M0, T1-4N1-3M0 (according to AJCC2009);
* No radiotherapy, chemotherapy or other treatments pre (post) surgery;
* PS ECOG 0-2;
* Life expectancy of more than 3 months;
* Hemoglobin (Hb) ≥ 9 g/dL • WBC ≥ 3 x 109/L, Neutrophils (ANC ) ≥ 1.5 x 109/L • platelet count (Pt) ≥ 100 x 109/L • Hepatic function: ALAT and ASAT < 2.5 x ULN, TBIL< 1.5 x ULN • Renal function: creatinine < 1.5 x ULN
* No immuno-deficiency;
* Use of an effective contraceptive for adults to prevent pregnancy.

Exclusion Criteria:

* Complete esophageal obstruction after surgery, Esophageal perforation, Haematemesis;
* Other malignant tumors, except for skin basal cell carcinoma, or cervical carcinoma in situ, who survived with no evidence disease for over 3 years;
* Participation in other interventional clinical trials within 30 days;
* Pregnant or breast-feeding women or people during the birth-period who refused to take contraceptives;
* Drug addiction, Alcoholism or AIDS;
* Uncontrolled seizures or psychiatric diseases, loss of control over their own behavior;
* Unsuitable to be enrolled in the trial in the opinion of the investigators.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
Local control rate | 2 years

SECONDARY OUTCOMES:
overall survival | 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan Universtiy Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Shen J, Ai D, Chen Y, Liu Q, Deng J, Hao S, Zhang X, Zhang J, Zhang Y, Chu L, Sun Y, Zhang Y, Xiang J, Miao L, Chen H, Zhu H, Zhao K. Postoperative chemoradiotherapy for esophageal squamous cell Carcinoma: Results from ESO-Shanghai 17 and joint analyses for phase II clinical trials. Clin Transl Radiat Oncol. 2025 Nov 21;57:101073. doi: 10.1016/j.ctro.2025.101073. eCollection 2026 Mar. PMID 41531940
- [Derived] Ai D, Chen Y, Liu Q, Deng J, Zhang X, Zhang J, Chu L, Shen J, Ma L, Zhang Y, Chen H, Miao L, Zhao K, Xiang J. Extensive clinical target volume in postoperative chemoradiotherapy for esophageal squamous cell carcinoma: a phase II clinical trial (ESO-Shanghai 9). Radiat Oncol. 2023 Feb 7;18(1):26. doi: 10.1186/s13014-023-02211-w. PMID 36750858